CLINICAL TRIAL: NCT00864513
Title: A Phase II Study of Pemetrexed as Second-Line Treatment in Patients With Pancreatic Cancer Progressing Despite Therapy With Gemcitabine
Brief Title: Study of Pemetrexed for Second-Line Pancreas Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: At interim analysis the study did not meet the response criteria to continue
Sponsor: Georgetown University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jimmy Hwang, Principal Investigator, Georgetown University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2007022; 2007-022
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Pancreas Cancer
Keywords: pancreas; metastatic; recurrent
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemotherapy (Experimental): pemetrexed
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — pemetrexed 500 mg/m2 IV day 1 of each 21 day cycle until disease progression or unacceptable toxicity for a maximum of 8 cycles
  Other Names: Alimta; LY231514; NSC# 698037

SUMMARY:
This study is for patients with pancreatic cancer that has grown and/or spread after having previously received the standard chemotherapy drug called gemcitabine.

In this study a drug called pemetrexed is being tested. This drug is approved by the FDA for use in lung cancer and mesothelioma. The purpose of this study is to see if pemetrexed keeps pancreas cancer that has grown and/or spread after gemcitabine from growing. Subjects will receive pemetrexed IV once every 21 days until disease progression or unacceptable side effects occur.

DETAILED DESCRIPTION:
This is an open label Phase II trial using pemetrexed as second-line treatment in patients with advanced pancreatic cancer progressing within six months of prior gemcitabine-based therapy. Subjects will receive pemetrexed 500 mg/m2 IV every 21 days until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas
* Prior treatment for distant or locally advanced disease with gemcitabine-based therapy
* Measurable or evaluable disease
* ECOG performance status 0-2
* Adequate hematological parameters
* Adequate baseline liver function
* At least 28 days from any major surgery
* At least 2 weeks from the last radiation treatment
* Must have recovered from reversible toxicities of prior chemotherapy
* Must be able to discontinue any nonsteroidal anti-inflammatory medications
* Must be willing to receive intramuscular vitamin B12 shots and take oral folate supplements

Exclusion Criteria:

* Any prior treatment with pemetrexed
* More than one prior chemotherapy regimen
* HIV positive on antiretroviral therapy
* Pregnant or lactating
* Prior organ allograft
* On concurrent antitumor therapy including radiation therapy or other chemotherapies
* Creatinine clearance 45 ml/min or less
* Absolute neutrophil count < 1500
* Platelets < 75,000
* Bilirubin > 1.5 times the upper limit of normal
* Transaminases > 3 times the upper limit of normal except in known liver metastasis wherein they may be </= 5 times upper limit of normal
* Clinically significant ascites or pleural effusion that cannot be drained
* Any medical or psychiatric condition that may interfere with the ability to comply with protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy J Hwang, M.D., Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital/Lombardi Cancer Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 12/2007 to 3/2009 17 patients were enrolled; 2 of which did not receive any treatment.
Groups:
- Chemotherapy: Subjects will be treated with pemetrexed 500 mg/m2 IV once every 21 days. They are also premdicated with dexamethasone 4 mg po BID on the day before, of and after chemotherapy. They will start folic acid 350-1000mcg by mouth daily, 5-7 days before starting study therapy. They will also receive a 1000 mcg IM injeciton of vitamin B12 1-2 weeks before study drug, and eveyr 9 weeks thereafter, until 3 weeks after the last dose of study treatment
Period: Overall Study
Arm/Group | Chemotherapy
Started | 15
Completed | 12
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Number of days from first dose of study treatment until the date of progression, as measured by worsening disease (new site of disease, or increase in existing disease) or death.
Time Frame: 6 months after last patient enrolled
Measure: Median (Full Range); unit: days
Arm/Group | Chemotherapy
Number analyzed (Participants) | 15
days | 59 [26 to 241]

2. Secondary Outcome: Objective Response
Description: Evaluation of tumor extent by CT scans, according to RECIST criteria (a 20% decrease in the sum of the longest unidimensional measurements of existing disease), version 1.0
Time Frame: Within two months of the completion of the last dose of chemotherapy
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 12
participants | 0

3. Secondary Outcome: CA 19-9 Response
Description: CA 19-9 was evaluatd every three weeks, before the next study treatment. Approximately 30% of patients are not expected to have detectable CA 19-9, based on Lews-Y antigen. CA 19-9 response is defined as more than 50% decrease from baseline.
Time Frame: Within two months of the last dose of chemotherapy
Population: Only 10 patients had elevated CA 19-9 at the start of therapy, and were therefore analyzable for this endpoint
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 10
participants | 2

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Toxicity by National Cancer Institute Common Toxicity Criteria Adverse Event Version 3.0
Time Frame: 30 days after last dose of study drug
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 15
participants | 2

ADVERSE EVENTS:
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=15)
neutropenia (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
study was closed at interim analysis so only 12 subjects were evaluable for response, 15 subjects received treatment and were evaluable for adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes